CLINICAL TRIAL: NCT06507982
Title: Comparison of Electronic Apex Locator and Simultaneous Working Length Detection Methods With Radiological Method in Terms of Postoperative Pain
Brief Title: Simultaneous Working Length Detection Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Seyda Ersahan, DDS, PhD, Principal Investigator, Clinical Associate Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 491
Record Dates: First submitted 2024-05-16; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Irreversible Pulpitis; Root Canal Treatment
Keywords: working length; irreversible pulpitis; apex locator; radiography; simultaneous measurement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization process of the patients participating in the study into groups was carried out by two endodontists (M.U. and S.E.) working in the unit where the research was conducted. Patients who met the inclusion criteria were randomly assigned to one of 3 groups. Additionally, patients requiring RCT for more than one tooth were randomly assigned to groups to ensure objectivity and maintain equal sample size.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Electronic working length method (Experimental): Electronic apex locator was used
  Interventions: Device: EWL
- Simultaneous working length method (Experimental): Working length was determined by EAL and then during root canal preparation, an endodontic motor using simultaneous working length control was selected
  Interventions: Device: SWL
- Radiologic working length method (Placebo Comparator): 30 patients in whom the radiologic working length (RWL) method. In this method, periapical radiographs were taken.
  Interventions: Device: RWL

INTERVENTIONS:
Device: EWL — the working length determination with EAL method
  Arms: Electronic working length method
Device: SWL — In this method, an endodontic motor with a built-in EAL that provides continuous feedback during root canal instrumentation and allows clinicians to make real-time adjustments to the WL. Thus, it provides continuous feedback, allowing the clinician to make real-time adjustments. The motor of devices using this method has automatic apical reverse and automatic apical stop operation. In this way, when the tip of the file reaches the apical foramen, the file safely reverses and stops rotating.
  Arms: Simultaneous working length method
Device: RWL — Radiographic method was used for determining the working length
  Arms: Radiologic working length method

SUMMARY:
Precise knowledge of the apical construction, which determines the end of the area for canal preparation and filling, is essential for the success of root canal treatment and the management of postoperative pain. For this purpose, devices based on various methods that determine the working length are used. However, it is still controversial which method provides the most accurate measurements.In this study, the compatibility of the electronic apex locator (EAL) and simultaneous working length determination (SWL) methods in single-root teeth was investigated in comparison with the radiographic working length determination method (RWL) method, and to determine which one produced more effective results in terms of postoperative pain.A hundred patients applied for endodontic treatment with a diagnosis of irreversible pulpitis (IP) were included in the study, which was planned as a single-center prospective cohort. Patients were divided into three groups according to the method used to determine the root canal working length (WL). 35 patients in whom the WL with EAL method (EWL) was used were included in Group 1; 35 patients in whom the SWL method was used were included in Group 2; 30 patients in whom the RWL method was used were assigned to Group 3. Patient groups were randomly selected from people similar in age and gender. Age, gender, simplified oral hygiene index (OHI-S), oral and dental examinations and Visual Analogue Scale (VAS) results of all participants were recorded.

DETAILED DESCRIPTION:
Devices that apply various methods to determine the root canal working length have been developed. The simultaneous working length determination is a newer development that allows clinicians to clean and shape root canals while monitoring the file's position inside the canal using dynamic feedback from EAL. In this method, an endodontic motor with a built-in EAL that provides continuous feedback during root canal instrumentation and allows clinicians to make real-time adjustments to the WL. Thus, it provides continuous feedback, allowing the clinician to make real-time adjustments. The motor of devices using this method has automatic apical reverse and automatic apical stop operation. In this way, when the tip of the file reaches the apical foramen, the file safely reverses and stops rotating. Thereby, SWL method reduces the risk of over- instrumentation. In this study, planned in the light of the above information, the aim of this study was to investigate the compatibility of the EWL and SWL methods in single-root teeth, in comparison with the RWL method, and to determine which one produces more effective results in terms of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of irreversible pulpitis Clinical indication for root canal treatment Able to come for follow-ups

Exclusion Criteria:

cardiovascular disease antibiotic or antienflammatuary drug usage during last 3 months excess coronal structure damage for rubber dam placement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain evaluation by VAS scale | Baseline, 24 hour postoperatively, 48hour postoperatively, 72 hour postoperatively, Day 3 and Day 7
  during first week after root canal treatment, postoperative pain was evaluated. From start of endodontic treatment up to 1 week, pain was evaluated using VAS scale VAS scale was used, which has 1 to 10 number Number 10 in VAS indicates severe pain, while 0 indicates no pain

CONTACTS AND LOCATIONS:
Overall Officials: Emine Guzel, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Upon request from the authors with a reasonable request, our data will be made open
Supporting Information: Study Protocol, SAP
Time Frame: After the acceptance of our study
Access Criteria: Our data will be shared via email